CLINICAL TRIAL: NCT01916395
Title: Comparison of Treximet and Imitrex as They Affect the Levels of Inflammatory Markers When the Patient is Actively Having a Migraine Headache.
Brief Title: Comparison of Treximet & Imitrex as They Affect the Levels of Inflammatory Markers When the Patient is Actively Having a Migraine Headache
Status: Completed | Type: Observational
Sponsor: Gary E. Ruoff, M.D. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Gary E. Ruoff, M.D., Director of Clinical Research, Westside Family Medical Center, P.C.
Organization: Westside Family Medical Center, P.C. (Other)
Other Study IDs: GR10
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2009-12

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; sumatriptan-naproxen

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imitrex and Treximet: Imitrex 100mg as needed Treximet 85/500mg
  Interventions: Drug: sumatriptan and Treximet

INTERVENTIONS:
Drug: sumatriptan and Treximet — sumatriptan 100mg tablet when migraine is moderate or severe in intensity. Treximet 85/500mg tablet when migraine is moderate or severe in intensity.
  Other Names: Imitrex 100mg; Treximet 85/500mg

SUMMARY:
The primary objective is to determine whether inflammatory markers, such as C-Reactive Protein (CRP), Calcitonin Gene-Related Peptide (CGRP), Vasoactive Intestinal Polypeptide (VIP), or Substance P (SP) are reduced in patients having a migraine headache when treated with Imitrex or Treximet.

The secondary objective is to determine the effects of Imitrex and Treximet on C-Reactive Protein (CRP) in patients with active migraine headaches.

DETAILED DESCRIPTION:
Migraine is a neurovascular process involving the brain and related structures. Neuroinflammatory substances such as CRP, CGRP, VIP, SP, and prostaglandins are liberated during the migraine. Elevation of these markers may be associated with other conditions which contain an inflammatory component such as coronary artery disease. VIP is an inflammation and pain transmission, and thus are markers of sensory nociceptive neurons.

During this study, the subjects will have the following inflammation markers analyzed: C-Reactive Protein (CRP), Calcitonin Gene-Related Peptide (CGRP), Vasoactive Intestinal Polypeptide (VIP), and Substance P (SP).

ELIGIBILITY:
Inclusion Criteria:

* Subject must sign an informed consent
* Males and females 18 - 65 years of age
* Have episodic migraine headaches
* Patients to satisfy the diagnosis of migraine headaches with aura, without aura or mixed
* Must be able to differentiate migraine headaches from other headaches
* Diagnosis of migraines for at least 6 months

Exclusion Criteria:

* Any medical condition, in the opinion of the investigator, that would make the subject unsuitable for enrollment
* Basilar or hemiplegic migraine headaches
* Pregnant woman or a nursing mother
* History (within 1 year) or current evidence of grug or alcohol abuse
* More than 15 migraine headaches per month
* Chronic daily headache
* Chronic use of NonSteroidalAntiInglammatoryDrugs
* Current participation in a research study or within the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients with migraine headaches.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The outcome will be to determine whether inflammatory markers are reduced in patients having a migraine when treated with Imitrex 100mg or Treximet. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary E Ruoff, MD, Principal Investigator — Family Practice
Locations (1):
- Westside Family Medical Center, PC, Kalamazoo, Michigan, United States